CLINICAL TRIAL: NCT03401320
Title: A Phase I, Open Label, Dose Escalation Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Single Intramuscular Injections of Letrozole ISM® at Different Strengths in Voluntary Healthy Post Menopausal Women (LISA-1)
Brief Title: Evaluation of IM Letrozole ISM® Pharmacokinetics, Safety, and Tolerability in Healthy Post-menopausal Women (LISA-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ROV-LET-2017-01; LISA-1 (Other: Rovi)
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: pharmacokinetics; letrozole
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: Phase I, open label, sequential, single ascending dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: Letrozole ISM 50 mg (Experimental): 14 oral doses of 2.5 mg Femara (once daily) + single IM injection of 50 mg Letrozole ISM
  Interventions: Drug: Letrozole ISM
- Cohort 2: Letrozole ISM 100 mg (Experimental): 14 oral doses of 2.5 mg Femara (once daily) + single IM injection of 100 mg Letrozole ISM
  Interventions: Drug: Letrozole ISM
- Cohort 3: Letrozole ISM 200 mg (Experimental): 14 oral doses of 2.5 mg Femara (once daily) + single IM injection of 200 mg Letrozole ISM
  Interventions: Drug: Letrozole ISM
- Cohort 4: Letrozole ISM 400 mg (Experimental): 14 oral doses of 2.5 mg Femara (once daily) + single IM injection of 400 mg Letrozole ISM
  Interventions: Drug: Letrozole ISM

INTERVENTIONS:
Drug: Letrozole ISM — 2.5 mg Femara + single IM injection of 50-400 mg Letrozole ISM
  Other Names: Femara; 4,4'-(1H- 1,2,4-Triazol-1-ylmethylene)dibenzonitrile

SUMMARY:
This is a Phase I, open label, dose escalation study designed to evaluate the pharmacokinetics, safety, and tolerability of single intramuscular injections of Letrozole ISM® at different strengths in voluntary healthy post menopausal women

DETAILED DESCRIPTION:
The objective of this study is to assess the pharmacokinetic profile of a single ascending doses of Letrozole ISM® (Rovi), and secondly, to evaluate safety and tolerability of single ascending doses of Letrozole ISM, measure estrogen levels, and characterize oral letrozole pharmacokinetic profile to be used in subsequent comparison to Letrozole ISM.

The study will be carried out in healthy post-menopausal women who satisfy inclusion and exclusion criteria.

The study consists of 3 treatment periods (TP) (TP1, TP2 and TP3) preceding by 2 Screening Periods (one for TP1 and one for TP3). In TP1, each subject will sequentially receive 1 dose daily of oral Femara (EU sourced) over a period of 14 days followed by a single intramuscular (IM) dose of Letrozole ISM (after a washout period) in TP2. Ascending doses of Letrozole ISM will be given sequentially to four Cohorts (1, 2, 3, and 4) [NOTE: Cohorts 3 and 4 were not finally performed because the Safety Review Committee considered it was not necessary for the achieving the objectives of the study] . All subjects who will finalize TP2 and fulfil the eligibility criteria will be offered to participate in TP3. The purpose is to have, at least, a minimum of 12 subjects receiving one oral daily dose of Femara (US sourced) 2.5 mg QD for a period of 14 days, to provide a complete pharmacokinetic (PK)/pharmacodynamic (PD) face-to-face comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy post-menopausal women, ≥ 18 and ≤ 75 years of age, who have achieved complete menopause, either natural or surgical, and amenorrhea, and have not been on hormone replacement therapy in the last 3 months.
2. Post-menopausal subjects should have absence of menses for 1 year, and oophorectomized subjects should have absence of menses for at least 6 weeks. For oophorectomized subjects and subjects who have had a hysterectomy, a surgical pathology report documenting the absence of malignant disease is required. In addition, for oophorectomized subjects an operative report documenting bilateral oophorectomy is required.
3. Baseline follicle-stimulating hormone (FSH) and 17β-estradiol plasma levels should be consistent with the post-menopausal status of the subject (FSH ≥ 40 mIU/mL; 17β-estradiol ≤ 31 pg/mL), confirmed at least 48 hours prior to dosing.
4. Weight of ≥ 50 kg and a BMI ≥ 19 and ≤ 39 kg/m2.
5. Subjects will be in good health, as determined by medical history, physical examination, vital signs assessments (pulse rate, systolic and diastolic blood pressure, and temperature), clinical laboratory evaluations, and 12-lead ECG. Minor deviations outside the reference ranges will be acceptable, if deemed not clinically significant by the investigator.
6. Subjects who have not had a mammogram within the last 12 months (documentation required) must be willing to have one performed.
7. Subjects with an intact uterus and cervix who have not had a Papanicolaou (pap) smear test within the last 6 months (documentation required) must be willing to have one performed.
8. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.
9. Subjects should be able to communicate with clinic staff.

Exclusion Criteria:

1. Subjects who have a history of allergy or hypersensitivity to letrozole or any of the inactive ingredients in the last 3 months.
2. Subjects who have a history of galactose intolerance, severe hereditary lactase deficiency glucose-galactose malabsorption.
3. Subjects who have used estrogen or progesterone hormone replacement therapy, thyroid replacement therapy, oral contraceptives, androgens, luteinizing hormone (LH) releasing hormone analogs, prolactin inhibitors, or antiandrogens within 3 months prior to Screening.
4. Subjects who have regularly taken foods or food supplements that contain high levels of Isoflavinoids, including soybean, soymilk, soynuts, chickpeas, alfalfa, fava beans, kudzu, miso and tofu in the 14 days prior to dosing (Treatment Period 1).

   4.1. The investigator and medical monitor will determine on a case-by-case basis if a subject who intakes food or food supplements containing Isoflavinoids is eligible to participate in the study.
5. Subjects who have used:

   5.1. Any medications including St. John's wort, known to be potent or moderate inducers of CYP P450 3A4 in the 3 weeks prior to dosing (Treatment Period 1).

   5.2. Any medications or products known to be potent or moderate inhibitors of CYP P450 3A4 (e.g. grapefruit juice) in the 7 days prior to dosing on Treatment Period 1.
6. Any prescribed preparations within 14 days prior to dosing (Treatment Period 1), unless in the opinion of the investigator (or designee) the medication will not interfere with the study procedures or compromise safety.
7. Any non-prescribed systemic or topical medications within 7 days of dosing (Treatment Period 1) unless in the opinion of the investigator (or designee) the medication will not interfere with the study procedures or compromise safety. Vitamins and minerals including the use of calcium and/or vitamin D for osteoporosis prevention are allowed.
8. Subjects who have been diagnosed with osteoporosis (previously or results from screening DEXA for this study with a T score < -2.5). Subjects with osteopenia (with the T-score between -1 and -2.5) will be allowed to participate in this study.

   8.1. Subjects who are not on a stable dose of long- or short-acting bisphosphonates therapy for at least 3 months prior to Screening.

   8.2. Subjects who are on raloxifene therapy.
9. Subjects who have an abnormality in heart rate, blood pressure, or temperature at Screening and prior to first dose (Treatment Period 1) that in the opinion of the investigator increases the risk of participating in the study. Resting SBP must be ≤ 150mmHg and resting DBP ≤ 95 mmHg.
10. Subjects who have an abnormality in the 12-lead ECG at Screening and prior to first dose (Treatment Period 1) that in the opinion of the Investigator increases the risk of participating in the study.
11. Subjects who have any clinically significant abnormal physical examination finding.
12. Subjects who have any clinically significant abnormal laboratory safety findings at Screening or Check-in, upon repeat testing, as determined by the investigator (1 repeat assessment is acceptable).

    12.1. Subjects who have ALT or AST >1.5 × ULN. For subjects with elevated total bilirubin, direct and indirect bilirubin will be evaluated.

    12.2. Subjects with elevated cholesterol or triglyceride levels above the ULN must be determined by the Investigator to be not clinically significant.
13. Subjects who have relevant diseases or clinically significant abnormal relevant findings at Screening, as determined by medical history, physical examination, laboratory, ECG, DEXA, and breast and pelvic examination.
14. Subjects who have history of any significant chronic disease, such as but not limited to: thrombotic disorders, coronary artery or cerebrovascular disease, liver, kidney or gallbladder dysfunction/disorder(s), diabetes or any other endocrine disease, estrogen dependent neoplasia, post-menopausal uterine bleeding, or endometrial hyperplasia. Subjects with cholecystectomy will be permitted if no medical sequelae post-surgery.
15. History of cancer within the past 5 years with the exception of non-melanoma skin cancer.
16. Subjects who have a history of drug-dependence, and recent history of alcoholism or abuse of alcohol.
17. Subjects who have a positive result for hepatitis B surface antigen (HBsAg), hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus (HIV) antibodies.
18. Subjects with a positive drugs of abuse screen or alcohol breath test at Screening (urine will be screened for the presence of the following: amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiates, phencyclidine, and methadone).
19. Subjects with a history of, or difficulty of, access to veins for venipuncture.
20. Subjects who have donated blood in the 30 days prior to first dose (Treatment Period 1).
21. Subjects who have received blood products within 2 months prior to Screening.
22. Subjects who have received a drug in research or have participated in other clinical trials within 30 days, or 5 half-lives (whichever is longer) prior to dosing (Treatment Period 1).
23. Subjects who have previously taken part in or have withdrawn from this study. (Subjects who have been screened for but not included in a cohort or subjects who dropped out from screening in a previous cohort for non-medical reasons may be eligible to be included in subsequent cohorts.)
24. Any other unspecified reason that, in the opinion of the investigator (or designee) or Sponsor, makes the subject unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
λz | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Terminal phase elimination rate constant
Cmax | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Maximum observed plasma concentration
Cmax/D | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Dose-normalized Maximum observed plasma concentration
tmax | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Time to maximum observed concentration
tlag | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Lag time before observation of quantifiable concentrations in plasma
t½ | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Terminal elimination half life
AUC∞ | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Area under the concentration time curve from time zero extrapolated to infinity
AUC∞/D | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Dose-normalized AUC∞
AUCextrap | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Percentage of AUC∞ obtained by extrapolation
AUClast | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Area under the concentration time curve from time zero up to the last quantifiable concentration
Vz/F | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Apparent volume of distribution during terminal phase after extravascular dosing
CL/F | Following single intramuscular administration of Letrozole ISM (Period 2, Day 1)
  Apparent systemic clearance after extravascular dosing

SECONDARY OUTCOMES:
λz | Following multiple oral administrations of Femara (Period 1, Day 14)
  Terminal phase elimination rate constant
Cav | Following multiple oral administrations of Femara (Period 1, Day 14)
  Average plasma concentration over a dosing interval
Cmin,ss | Following multiple oral administrations of Femara (Period 1, Day 14)
  Minimum observed plasma concentration at steady state
Cmax,ss | Following multiple oral administrations of Femara (Period 1, Day 14)
  Maximum observed plasma concentration at steady state
tmax | Following multiple oral administrations of Femara (Period 1, Day 14)
  Time to maximum observed concentration
t½ | Following multiple oral administrations of Femara (Period 1, Day 14)
  Terminal elimination half life
AUCτ | Following multiple oral administrations of Femara (Period 1, Day 14)
  Area under the concentration time curve over a dosing interval
Vz/F | Following multiple oral administrations of Femara (Period 1, Day 14)
  Apparent volume of distribution during terminal phase after extravascular dosing
CLss/F | Following multiple oral administrations of Femara (Period 1, Day 14)
  Apparent systemic clearance after extravascular dosing at steady state
Hormones levels | From date of screening to follow-up visit, assessed up to 50 weeks
  The dose response relationship between doses letrozole and some hormones levels
AEs | From date of screening to follow-up visit, assessed up to 50 weeks
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martínez, MD, Study Director — Laboratorios Farmaceuticos Rovi, S.A.
Locations (1):
- Investigational Site Number 42001, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No